CLINICAL TRIAL: NCT03546517
Title: Effectiveness of Dry Needling (DNHS Technique) in Patients With Chronic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad San Jorge (Other)
Responsible Party: Principal Investigator, Pablo Herrero Gallego, Head of iPhysio Research Group, San Jorge University, Universidad San Jorge
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DNHS_stroke
Record Dates: First submitted 2018-04-20; First posted 2018-06-06 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Stroke; Spasticity
Keywords: myofascial trigger point; dry needling; spasticity; stroke
MeSH Terms: conditions — Stroke; Muscle Spasticity | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients and assessor are blinded but the physiotherapist giving the treatment is not blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention with DNHS technique (Experimental): Dry needling of biceps brachii, brachialis, flexor digitorum superficialis and flexor digitorum profundus, triceps brachialis, extensor digitorum and adductor pollicis
  Interventions: Other: Dry Needling
- Sham Dry Needling (Sham Comparator): Sham Dry needling of biceps brachii, brachialis, flexor digitorum superficialis and flexor digitorum profundus, triceps brachialis, extensor digitorum and adductor pollicis
  Interventions: Other: Sham Dry Needling

INTERVENTIONS:
Other: Dry Needling — Dry needling of biceps brachii, brachialis, flexor digitorum superficialis and flexor digitorum profundus, triceps brachialis, extensor digitorum and adductor pollicis
  Other Names: DNHS technique
  Arms: Intervention with DNHS technique
Other: Sham Dry Needling — Sham Dry needling of biceps brachii, brachialis, flexor digitorum superficialis and flexor digitorum profundus, triceps brachialis, extensor digitorum and adductor pollicis
  Arms: Sham Dry Needling

SUMMARY:
Study hypothesis:

The DNHS technique, performed via one session of deep dry needling of myofascial trigger points applied to the biceps brachii, brachialis, flexor digitorum superficialis, flexor digitorum profundus, triceps brachii, extensor digitorum and adductor pollicis muscle is effective for decreasing spasticity and muscle stiffness (both of which are components of hypertonia) as well as for improving the upper limb function of the previously described muscles in patients with chronic cerebral vascular accident (CVA), assessed both post-intervention and after 15 days.

General aims

To analyse the immediate therapeutic effect of the DNHS technique and the effect at 15 days follow-up, for the following variables:

* Spasticity
* Muscle stiffness
* Upper limb function
* Patient perceived quality of life

Materials and methods Population: patients from the province of Zaragoza (Spain) diagnosed with a haemorrhagic or ischemic CVA by a neurologist.

Recruitment strategy: recruitment will take place via the Stroke Association in Aragon (AIDA) [Aragon Stroke Association] in the province of Zaragoza, Spain, seeing as the greater proportion of patients who have suffered a stroke and are in the chronic stage of the illness go to this centre to receive treatment. Thus, this avoids patients having to travel elsewhere for the study. Furthermore, in the case of patients who wish to participate in the study after having received information via third persons or via other means and who are not members of the Association or do not attend the centre on a regular basis, the Association AIDA has offered to allow these people to attend for free, making its facilities available and supporting the development of this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been diagnosed with a haemorrhagic or ischemic CVA by a neurologist.
* Cognitive level: minimental state examination (MMSE) ≥ 27 points. All patients must have a good cognitive level in order to ensure that they are able to communicate with the professionals involved in the study in order to understand the exercises and thus fulfil the objectives for participation.
* Presence of spasticity ≥1 according to the Modified Modified Ashworth Scale (MMAS) score during the flexion-extension movement of the wrist and elbow in at least one of the muscles of the upper limb evaluated.
* Age: between 30 - 90 years. In this range of age CVA's are more common, according to data from the Spanish Statistical Office.
* Evolution: over 6 months must have passed since the CVA episode. Most of the studies reviewed involve patients who are in the chronic stage of illness. This will ensure that the changes found are due to our intervention and not related to plasticity mechanisms occurring after the injury (this will be considered objectively by performing an assessment at baseline, which will be repeated 1 week later, immediately before and after the dry needling intervention).

Exclusion Criteria:

* Concomitance of degenerative illnesses which can alter the results.
* Presence of fixed contractures: 4 according to the MMAS score
* Suffering from epileptic fits that are not medically controlled.
* Fear of needles.
* No tolerance to pain caused by needling.
* Those unable to commit to attendance.
* Patients who have received treatment with Botulinum Toxin (BTX A) in the 6 months prior to their inclusion in this study, or those who received said medication or another during the study with the aim of decreasing spasticity.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-09-04 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Scale | Change between baseline (immediately before intervention) and post intervention (immediately after intervention). Change between baseline (immediately before intervention) and follow-up at 2 weeks after intervention
  Scale measuring Upper Limb Function in stroke patients. The motor and sensory assessments are scored on a three-point ordinal scale (0 -2) in which a higher score indicates superior results. The motor assessment measures voluntary limb movement and includes a subscale for the Upper Extremity (33 items; score range, 0-66). The sensory assessment measures limb sensation. Sensation is assessed as absent, impaired, or normal for light touch (two items each for Upper Extremity (UE) and Lower Extremity (LE); score range, 0-8) and proprioception (four items each for UE and LE; score range, 0-16) for a total sensory Fugl-Meyer (FM) score of 24. Fugl-Meyer Assessment (FMA) has shown to have an excellent intra and interrater reliability (0.89-0.99). The estimated minimal clinical important difference (MCID) of the UE-FM scores ranged from 4.25 to 7.25 points .

SECONDARY OUTCOMES:
Modified Modified Ashworth Scale | Change between baseline (immediately before intervention) and post intervention (immediately after intervention). Change between baseline (immediately before intervention) and follow-up at 2 weeks after intervention
  Scale measuring Spasticity/Hypertonia. This scale ranges from 0 to 4 points for each muscle assessed, where 0 is no hypertonia/spasticity and 4 is the highest hypertonia/spasticity.
Electromyography (EMG) | Change between baseline (immediately before intervention) and post intervention (immediately after intervention). Change between baseline (immediately before intervention) and follow-up at 2 weeks after intervention
  Neurophysiological measurements (electromyographic measurements). The amount of electrical activity will be measured quantitatively, from 0 to an undefined value (depending on every muscle´s activity)
Tonometry (measurement of muscle tone with a device) | Change between baseline (immediately before intervention) and post intervention (immediately after intervention). Change between baseline (immediately before intervention) and follow-up at 2 weeks after intervention
  Muscle stiffness or muscle tone. This device register different parameters like frequency, oscillation, etc that are related to tone, and start from 0 to an undefined number (depending on every muscle). It is a quantitative measurement.
Quality of Life (Euro QoL5D) | Change between baseline (immediately before intervention) and follow-up at 2 weeks after intervention
  Quality of Life. This scale measures quality of life. Description: This is a measure of self-reported health outcomes. It consists of two parts: a descriptive system (Part I) and a visual analogue scale (VAS) (Part II). Part I of the scale consists of 5 single-item dimensions including: mobility, self care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has a 3 point response scale, ranging from worst imaginable health state to best imaginable health state. Scoring/Interpretation: Descriptive data from the 5 dimensions of Part I can be used to generate a health-related quality of life profile for the subject. Part II is scored from 0 (worst health state imaginable) to 100 (best health state imaginable).

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad San Jorge, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No
Data will be available under request once it is published

REFERENCES:
- [Derived] Calvo S, Brandin-de la Cruz N, Jimenez-Sanchez C, Bravo-Esteban E, Herrero P. Effects of dry needling on function, hypertonia and quality of life in chronic stroke: a randomized clinical trial. Acupunct Med. 2022 Aug;40(4):312-321. doi: 10.1177/09645284211056347. Epub 2021 Dec 13. PMID 34894776